CLINICAL TRIAL: NCT01004263
Title: A Worldwide, Open Label, Clinical Trial to Examine the Long Term Safety and Tolerability of Rizatriptan in Pediatric Migraineurs for the Treatment of Migraine With or Without Aura
Brief Title: A Study to Evaluate the Safety and Tolerability of Rizatriptan for Long Term Treatment of Acute Migraine in Children and Adolescents (MK-0462-086 AM3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0462-086; 2009_680
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2022-02

CONDITIONS: Acute Migraine With or Without Aura in Adolescents
Keywords: acute migraine with or without aura in adolescents
MeSH Terms: interventions — rizatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rizatriptan (Experimental): Rizatriptan benzoate
  Interventions: Drug: rizatriptan benzoate

INTERVENTIONS:
Drug: rizatriptan benzoate — Single dose of 5 mg or 10 mg orally disintegrating tablet at onset of migraine attack
  Other Names: MK-0462; Maxalt

SUMMARY:
To provide long term safety data for rizatriptan in children and adolescents. The primary hypothesis of the study is that rizatriptan is well tolerated in the long term treatment of acute migraine in pediatric patients age 12-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 12 and 17 years of age inclusive at screening Visit 1
* Patient weighs at least 20 kg (44 pounds)
* Patient has had a history of unilateral or bilateral migraine headache with or without aura >6 months with ≥1 to ≤8 mild, moderate or severe migraine attacks per month in the 2 months prior to screening Visit 1
* Patient has a history of migraine defined by International Headache Society (IHS) migraine definitions
* The parent or guardian and patient agree to the patient's participation in the study as indicated by parental/guardian signature on the consent form and patient assent
* For patients taking migraine prophylactic medication, treatment regimen is stable and has been taken for at least 3 months prior to Visit 1

Exclusion Criteria:

* Patient is pregnant or breast-feeding, or is a female expecting to conceive within the projected duration of study participation
* Patient has a history of mild migraine attacks or migraines that resolve in less than 2 hours
* Patient has basilar or hemiplegic migraine headaches
* Patient has >15 headache-days per month OR has taken medication for acute headache on more than 10 days per month in any of the 3 months prior to screening
* Patient has uncontrolled high blood pressure, uncontrolled diabetes, human immunodeficiency virus (HIV), any cancer, or any other significant disease
* Patient has a history cardiovascular problems or stroke
* Patient has either demonstrated hypersensitivity to or experienced a serious adverse event in response to rizatriptan
* Patient has demonstrated hypersensitivity to or experienced a serious adverse event in response to 3 or more classes of drugs (over-the-counter and prescription)
* Patient did not experience satisfactory relief from migraine pain to prior treatment with 2 or more adequate courses of 5-hydroxytryptamine 1 (5HT1) agonists
* Patient has a recent history (within the past year) or current evidence of drug or alcohol abuse or is a "recreational user" of illicit drugs
* Patient is currently taking monoamine oxidase inhibitors, methysergide, or propranolol, and is unable to tolerate withdrawal of these medications for the intervals required
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of screening
* Patient is legally or mentally incapacitated

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 674 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hewitt DJ, Pearlman E, Hamalainen M, Lewis D, Connor KM, Michelson D, Ceesay P, Assaid C, Bachman R, Harper Mozley L, Dupre N, Strickler N, Mahoney E, Lines C, Ho TW. Long-term open-label safety study of rizatriptan acute treatment in pediatric migraineurs. Headache. 2013 Jan;53(1):104-117. doi: 10.1111/j.1526-4610.2012.02285.x. Epub 2012 Oct 18. PMID 23078588

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 674 patients met inclusion/exclusion criteria and were allocated study drug. Of these, 606 were treated with study drug.
Groups:
- Rizatriptan: Participants self-administered rizatriptan to treat up to 8 qualifying migraine headaches (mild, moderate, or severe pain intensity) per month, for up to 12 months. Rizatriptan dose, administered as a single oral tablet, was either 5 or 10 mg, based on participant weight (5 mg if <40 kg, 10 mg if ≥40 kg).
Period: Overall Study
Arm/Group | Rizatriptan
Started | 606 (Participants who took study drug)
Completed | 427
Not Completed | 179
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 58
Not completed — Protocol Violation | 10
Not completed — Lost to Follow-up | 64
Not completed — Lack of Efficacy | 13
Not completed — Pregnancy | 2
Not completed — Physician Decision | 15
Not completed — Lack of Qualifying Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rizatriptan
Number analyzed (Participants) | 606
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 372
  Male | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Within 24 Hours Post Any Dose
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration. Participants reported AEs in a diary and these were collected by the study site at visits at 1, 2, 3, 4, 6, 9, and 12 months after Screening visit. Participants with an AE occurring within 24 hours after any dose administered during the study are counted once in this summary.
Time Frame: Up to 24 hours post dose
Population: All enrolled participants who administered at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Rizatriptan
Number analyzed (Participants) | 606
participants | 322

2. Primary Outcome: Number of Participants With AEs Within 14 Days Post Any Dose
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration. Participants reported AEs in a diary and these were collected by the study site at visits at 1, 2, 3, 4, 6, 9, and 12 months after Screening visit. AEs were assessed in a phone contact 14 days after the last dose of study medication. Participants with an AE occurring within 14 days after any dose administered during the study are counted once in this summary.
Time Frame: Up to 14 days post dose
Population: All enrolled participants who administered at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Rizatriptan
Number analyzed (Participants) | 606
participants | 400

3. Secondary Outcome: Percentage of Participant's Migraine Attacks With Pain Freedom at 2 Hours Post Dose
Description: Pain intensity was assessed using a 5-Face Pain Scale ranging from 1=no pain to 5=very bad pain. Pain freedom (PF) was defined as a reduction in severity from a rating of 5, 4, 3 or 2 (mild, moderate or severe pain) before the dose to a rating of 1 (no pain) at 2 hours after dosing. Pain intensity ratings were reported in diaries returned at visits at 1, 2, 3, 4, 6, 9, and 12 months after Screening visit. PF at 2 hours was summarized as follows: the percentage of treated attacks with PF at 2 hours was calculated for each patient first, then the mean across all patients was calculated.
Time Frame: 2 hours post dose
Population: All participants who were enrolled and reported at least one treated migraine attack with at least one post treatment efficacy evaluation
Measure: Mean (Standard Deviation); unit: percentage of participant's attacks
Arm/Group | Rizatriptan
Number analyzed (Participants) | 603
percentage of participant's attacks | 46.3 (31.9)

4. Primary Outcome: Number of Participants Discontinued From Study Due to AEs Occurring Within 24 Hours Post Dose
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration. Participants who discontinued due to an AE occurring within 24 hours post dose are counted in this summary.
Time Frame: Up to 24 hours post dose
Population: All enrolled participants who administered at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Rizatriptan
Number analyzed (Participants) | 606
participants | 4

5. Primary Outcome: Number of Participants Discontinued From Study Due to AEs Occurring Within 14 Days Post Dose
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration. Participants who discontinued due to an AE occurring within 14 days post dose are counted in this summary.
Time Frame: Up to 14 days post dose
Population: All enrolled participants who administered at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Rizatriptan
Number analyzed (Participants) | 606
participants | 14

ADVERSE EVENTS:
Time Frame: Up to 12 months after start of study drug administration
Description: AE tables include all enrolled participants who administered at least one dose of study medication
Arm/Group | Rizatriptan
Serious Adverse Events (participants affected / at risk) | 22/606
Other Adverse Events (participants affected / at risk) | 284/606
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rizatriptan (N=606)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (2)
Appendicitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Suicide attempt (Psychiatric disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rizatriptan (N=606)
Nausea (Gastrointestinal disorders) | 40 (77)
Fatigue (General disorders) | 33 (111)
Nasopharyngitis (Infections and infestations) | 47 (56)
Upper respiratory tract infection (Infections and infestations) | 31 (33)
Accidental overdose (Injury, poisoning and procedural complications) | 148 (216)
Dizziness (Nervous system disorders) | 52 (94)
Somnolence (Nervous system disorders) | 44 (123)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to delay publication of study results until Food and Drug Administration (FDA) grants pediatric exclusivity on the study drug. Investigator may publish results for his/her study site after primary publication of results of entire multicenter trial. Sponsor must be able to review all proposed results communications regarding study 60 days prior to submission for publication/presentation. Information identified by the Sponsor as confidential must be deleted prior to submission.